CLINICAL TRIAL: NCT01276041
Title: Paclitaxel, Trastuzumab, and Pertuzumab in the Treatment of Metastatic HER2-Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-142
Record Dates: First submitted 2011-01-06; First posted 2011-01-13 (Estimated); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: MAB 2C4 (PERTUZUMAB); MAB HER 2 (HERCEPTIN) (TRASTUZUMAB); TAXOL (PACLITAXEL); 10-142; Stage IV HER2 (+) breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab; Paclitaxel

ARMS (1):
- pertuzumab in combination with trastuzumab and paclitaxel (Experimental): This is a phase II study of pertuzumab in combination with trastuzumab and paclitaxel for the treatment of patients with Stage IV HER2 (+) breast cancer.
  Interventions: Drug: pertuzumab in combination with trastuzumab and paclitaxel

INTERVENTIONS:
Drug: pertuzumab in combination with trastuzumab and paclitaxel — The regimen will consist of paclitaxel (80 mg/m2) weekly + trastuzumab every 3 weeks (8 mg/kg loading dose → 6 mg/kg every 3 weeks) + pertuzumab every 3 weeks (840 mg as a loading dose → 420 mg), all given intravenously (IV). Patients may be given trastuzumab weekly in lieu of every 3 weeks (4 mg/kg loading dose → 2 mg/kg every 3 weeks). Patients will be on treatment until progression of disease.

SUMMARY:
The purpose of this study is to see if a combination of drugs can help to treat this type of cancer. One drug is a chemotherapy agent called paclitaxel (Taxol®). Paclitaxel will be given every week through the vein. Although the weekly schedule of paclitaxel is not included in the label, the schedule and dose of weekly paclitaxel have been studied and have been proven to be more effective than an old standard schedule. The other two work against HER2. One is called trastuzumab (Herceptin®) and it is commonly given to women with early HER2 positive breast cancer or with advanced HER2 positive breast cancer that has spread to other parts of the body. Trastuzumab will be given through the vein every 3 weeks (or every week at the doctor's discretion). The third drug, pertuzumab, is an investigational drug. It has not been approved by the Food and Drug Administration. It has been given in studies to over 800 people. It has been effective in treating HER2 positive breast cancer. Pertuzumab will be given every 3 weeks through the vein. This study is looking at the effectiveness of these three drugs together.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Stage IV HER2 (+) breast cancer.
* Histologically documented HER2 (+) breast cancer as defined as IHC 3+ or FISH amplification of ≥ 2.0 of primary or metastatic site; results from the local lab are acceptable. (Optional tumor sample collection from primary or metastatic site may be obtained for HER2 testing at MSKCC).
* ECOG performance 0 -1 (Appendix A)
* 0-1 prior treatment in the metastatic setting (ie: hormone, chemotherapy, biologic, targeted agents). Prior anthracycline, paclitaxel, and trastuzumab in the adjuvant setting are allowed. If the patient has one trastuzumab-based treatment in the metastatic setting and is given a break (even intermittently) from the partner drug given with trastuzumab and is continued on trastuzumab alone, this would still be considered as one treatment. For example, if the patient was given paclitaxel + trastuzumab and was later continued on trastuzumab alone or then restarted on paclitaxel + trastuzumab (at the physician's discretion for any reason), the regimen paclitaxel + trastuzumab followed by trastuzumab alone (or followed by paclitaxel + trastuzumab again) may be considered as one treatment.
* Measurable or non-measurable disease. Measurable lesions are defined as those that can be measured accurately in at least one diameter, that is 20 mm using conventional imaging techniques (including incremental CT) or 10 mm using spiral CT equipment and a lymph node 15 mm along the short axis. Non-measurable lesions are all other lesions, including small lesions (longest diameter <10mm pathological a lymph nodes with 10 to less than 15mm along the short axis, bony metastases, leptomeningeal disease, ascites, pleural/pericardial effusions, inflammatory breast cancer, lymphangitis carcinomatosis, and heavily calcified and cystic/necrotic lesions.
* LVEF ≥ 50%
* Hematologic parameters: white blood cell (WBC) count of ≥ 3000/ul, absolute neutrophil count (ANC) ≥1500/ul, platelets ≥ 100,000/ul, hemoglobin ≥ 10.0 g/dl
* Non-hematologic parameters: bilirubin ≤ 1.5 mg/dl, AST/ALT ≤ 2.5 x upper limit of normal (ULN), alkaline phosphatase ≤ 5 x ULN.
* Creatinine ≤ 1.5 mg/dl
* Patients with stable and treated brain lesions of a duration of ≥ 2 months may be enrolled.

Exclusion Criteria:

* History of prior cardiac morbidities within 12 months (unstable angina, myocardial infarction, CHF, uncontrolled ventricular arrhythmias)
* Prior pertuzumab
* History of prior ≥ G 3 hypersensitivity (HSR) or any toxicity to trastuzumab that warranted permanent cessation of this antibody
* History of prior ≥ G 3 HSR or any toxicity to paclitaxel warranted permanent cessation of this chemotherapy
* > G 2 peripheral neuropathy
* Patients with a history of chronic hepatitis B or C should be excluded from the study as paclitaxel is potentially hepatotoxic
* Pregnant patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-01-05 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chau Dang, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pertuzumab in Combination With Trastuzumab and Paclitaxel
Started | 70
Completed | 67
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pertuzumab in Combination With Trastuzumab and Paclitaxel
Number analyzed (Participants) | 70
Age, Continuous [Median (Full Range); unit: years] | 52 [26 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 43
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Are Progression Free at 6 Months or Later.
Description: Patients who are considered progression-free at 6 months are deemed successes. Failures are those patients who progressed before the 6 month mark. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of partcipants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Paclitaxel
Number analyzed (Participants) | 70
percentage of partcipants | 86 [75 to 93]

2. Secondary Outcome: Number of Participants by Response Rate Using the RECIST Criteria (Version 1.1)
Description: Extent of disease evaluation will consist of a CT of chest and abdomen +/- pelvis. Bone scan and PET are optional. Every 4th cycle, this can be done within +/- 2 weeks. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.",
Time Frame: every 4th cycle CT of chest and abdomen +/- pelvis up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Paclitaxel
Number analyzed (Participants) | 70
Participants
  Complete Response | 15
  Partial Response | 27
  Stable Disease | 17
  Progression of Disease | 1
  Not Evaulable | 10

3. Secondary Outcome: Number of Participants Evaluated for Cardiac Safety
Description: We will also assess the LVEF at baseline and after every 4th cycle of treatment with an ECHO with a strain imaging analysis. When an ECHO cannot be done, a MUGA scan may be done.Patients who have surpassed the 6 month period may complete ECHO with strain imaging analysis or MUGA every 6 months +/- 1 month starting from the most recent ECHO scan date. This study will use the NCI Common Toxicity Criteria (CTC) AE version 4.0 for toxicity.
Time Frame: baseline and every 4th cycle of treatment up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Paclitaxel
Number analyzed (Participants) | 70
Participants | 70

4. Secondary Outcome: Number of Participants Evaluated With Toxicity
Description: This study will use the NCI Common Toxicity Criteria (CTC) AE version 4.0 for toxicity.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Paclitaxel
Number analyzed (Participants) | 70
Participants | 70

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Pertuzumab in Combination With Trastuzumab and Paclitaxel
All-Cause Mortality (participants affected / at risk) | 36/70
Serious Adverse Events (participants affected / at risk) | 18/70
Other Adverse Events (participants affected / at risk) | 67/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab in Combination With Trastuzumab and Paclitaxel (N=70)
Abdominal Pain (Gastrointestinal disorders) | 5
Alanine aminotransferase increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blurred vision (Eye disorders) | 1
Breast infection (Infections and infestations) | 1
Cardiac arrest (Cardiac disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 1
Death NOS (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Edema cerebral (Nervous system disorders) | 2
Edema limbs (General disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 2
Fatigue (General disorders) | 3
Fever (General disorders) | 3
Gait disturbance (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 3
Hematoma (Vascular disorders) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Hydrocephalus (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Infections and infestations - other, specify (Infections and infestations) | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Lipase increased (Investigations) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal & conn tissue disorder Other, spec (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Nervous system disorders - other, specify (Nervous system disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 2
Sepsis (Infections and infestations) | 1
Serum amylase increased (Investigations) | 1
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 3
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab in Combination With Trastuzumab and Paclitaxel (N=70)
Diarrhea (Gastrointestinal disorders) | 60
Fatigue (General disorders) | 62
Alopecia (Skin and subcutaneous tissue disorders) | 57
Peripheral neuropathy (Nervous system disorders) | 59
AST/ALT elevation (Investigations) | 51
Cough (Respiratory, thoracic and mediastinal disorders) | 43
Dry skin (Skin and subcutaneous tissue disorders) | 44
Arthralgia (Musculoskeletal and connective tissue disorders) | 42
Nausea (Gastrointestinal disorders) | 42
Acneiform rash (Skin and subcutaneous tissue disorders) | 38
Mucositis (Gastrointestinal disorders) | 37
Peripheral edema (General disorders) | 36
Hot flashes (Vascular disorders) | 36
Xerophthalmia (Eye disorders) | 33
Dyspepsia (Gastrointestinal disorders) | 30
Epiphora (Eye disorders) | 30
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 29
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28
Anorexia (Metabolism and nutrition disorders) | 28
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT01276041/Prot_SAP_000.pdf